CLINICAL TRIAL: NCT07225413
Title: Dose-Response Effects of Short-Term *Rhodiola Rosea* on Anaerobic Performance and Cognitive Function in Resistance-Trained Adults: A Randomized, Double-Blind, Placebo-Controlled Crossover Trial
Brief Title: Short-Term Rhodiola Rosea for Anaerobic Performance and Cognitive Function in Resistance-Trained Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacksonville State University (Other)
Responsible Party: Principal Investigator, Majid Koozehchian, PhD, Associate Professor of Kinesiology; Program Coordinator, Human Performance & Nutrition; Principal Investigator, Jacksonville State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: JSU-EPNL-2025-01
Record Dates: First submitted 2025-10-31; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
Keywords: Rhodiola rosea; Golden root; Adaptogen; Dietary supplements; Resistance training; Strength training; Anaerobic performance; Wingate test; Executive function; Stroop Color-Word Test; Sports performance; Cognitive performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No-Capsule Control (No Intervention): Participants complete a 7-day control period during which no capsules are administered. On day 7 they report to the lab for testing (bench press and leg press 1RM, third set to failure at 60% 1RM, Tendo power, 30-s Wingate, and Stroop Color-Word Test), plus HR/BP and RPE. This arm is always completed first to establish baseline performance.
- Placebo (Placebo Comparator): Participants ingest placebo capsules once daily for 7 days. On day 7, ~60 minutes after the final dose, they complete the same performance and cognitive testing battery (resistance exercises, Wingate, Stroop, HR/BP, RPE). This arm controls for expectancy and capsule intake.
  Interventions: Dietary Supplement: Placebo capsules
- Low-Dose Rhodiola rosea (Experimental): Participants ingest low-dose Rhodiola rosea (e.g., 200 mg/day) for 7 days. On day 7, ~60 minutes after dosing, they complete the laboratory testing session (bench/leg press 1RM and 60% to failure, Tendo power, 30-s Wingate, Stroop test, HR/BP, RPE) to determine whether short-term low-dose RR improves strength, muscular endurance, anaerobic performance, or executive function relative to control and placebo.
  Interventions: Dietary Supplement: Rhodiola rosea (low dose)
- High-Dose Rhodiola rosea (Experimental): Participants ingest high-dose Rhodiola rosea (e.g., 1,500 mg/day) for 7 days. On day 7, ~60 minutes after dosing, they perform the identical performance and cognitive testing battery. This arm allows for comparison of a higher RR dose with low-dose, placebo, and control groups to assess dose-response effects on resistance performance and Stroop outcomes.
  Interventions: Dietary Supplement: Rhodiola rosea (high dose)

INTERVENTIONS:
Dietary Supplement: Rhodiola rosea (low dose) — Participants will ingest a low-dose Rhodiola rosea extract (≈approximately 200 mg/day) once daily for 7 consecutive days. On day 7, ~60 minutes after the final dose, they will complete the exercise and cognitive testing battery (bench press, leg press, set to failure at 60% 1RM, Tendo power, 30-s Wingate, Stroop test, HR/BP, RPE). This intervention is used to determine whether short-term, lower-dose RR improves resistance performance and executive function compared with placebo and control.
  Other Names: Rhodiola rosea extract 200 mg
  Arms: Low-Dose Rhodiola rosea
Dietary Supplement: Rhodiola rosea (high dose) — Participants will ingest a high-dose Rhodiola rosea extract (≈approximately 1,500 mg/day) once daily for 7 consecutive days. On day 7, ~60 minutes after the final dose, they will complete the same performance and cognitive testing battery. This arm allows dose-response comparison with the low-dose RR, placebo, and no-capsule control conditions.
  Arms: High-Dose Rhodiola rosea
Dietary Supplement: Placebo capsules — Participants will ingest matching placebo capsules once daily for 7 days. On day 7, ~60 minutes after capsule ingestion, they will complete the full testing battery. This intervention controls for expectancy, capsule handling, and timing.
  Arms: Placebo

SUMMARY:
This study will evaluate whether 7 days of Rhodiola rosea (golden root) supplementation can improve resistance-exercise performance and cognitive function in resistance-trained men and women. Participants will complete four 7-day periods in a randomized, double-blind, crossover order: (1) no-capsule control, (2) placebo, (3) low-dose Rhodiola rosea, and (4) high-dose Rhodiola rosea. On day 7 of each period, they will report to the laboratory for performance testing that includes bench press and leg press 1-repetition maximum (1RM), a third set to failure at 60% 1RM, Tendo-derived mean and peak power, a 30-second Wingate test, and the paper-and-pencil Stroop Color-Word Test for executive function. Secondary outcomes include ratings of perceived exertion, readiness to perform (visual analog scale), and heart rate and blood pressure measured at rest and 1 minute after exercise. The central hypothesis is that short-term Rhodiola rosea, compared with control and placebo, will produce small but measurable improvements in strength, set-to-failure volume, and Stroop performance, with minimal changes in hemodynamics.

DETAILED DESCRIPTION:
Rationale: Rhodiola rosea is an adaptogenic plant extract that has shown modest, context-dependent effects on perception of effort, cognition, and exercise performance. Prior studies suggest that benefits may be more evident with acute or short-term administration; however, the results are heterogeneous. This study employs a within-subject approach in resistance-trained adults to minimize between-person variability and investigate potential dose-response effects over a short time frame.

Design overview: After screening and a familiarization visit, each participant completes four 7-day periods: (1) no-capsule control, (2) placebo, (3) low-dose RR, and (4) high-dose RR. Capsule periods are randomized and double-blind; the no-capsule control precedes capsule periods to avoid carryover of expectancy. Study staff, participants, and outcome assessors are blinded during capsule periods. On day 7 of each period, participants attend a single testing visit conducted under standardized conditions (time of day, pre-test instructions). Short-latency effects are targeted by scheduling capsule ingestion approximately 60 minutes before testing during capsule periods.

Intervention: Low- and high-dose RR are provided in identical-appearing capsules. Placebo capsules contain inert filler. Product identity, dose, and lot information are recorded in the Intervention section of the record. Capsule count and participant logs monitor adherence.

Standardization and compliance: Participants are asked to maintain their habitual training and diet and to refrain from using additional ergogenic aids for a period of 7 days. They record total energy and macronutrients for the three days before each testing day. Testing sessions follow a consistent order of tasks established during the familiarization phase. Resting vital signs are obtained after a seated rest; post-exercise measures are obtained 1 minute after completion of designated tasks.

Population: Resistance-trained adults (men and women) who meet eligibility criteria and provide informed consent. Additional eligibility details are specified in the Eligibility section of the record. The female hormonal status/menstrual phases are documented when available to aid in interpretation.

Data handling and analysis (overview): The primary analyses compare conditions within participants using linear mixed-effects models, with participant as a random effect and fixed terms for condition and period. Additional prespecified covariates (e.g., sex, pre-visit dietary intake) may also be included. Order and carryover are evaluated as appropriate. Missing data are handled using model-based methods consistent with the statistical plan.

Safety: Adverse events are monitored throughout each period, with procedures for reporting to the IRB per institutional policy.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-40 years old
* ≥2 years of consistent resistance training, including bench press and leg press/squat
* Able to complete all four 7-day conditions and Day-7 testing in a crossover design
* Willing to abstain from other performance supplements during the study
* Provided written informed consent

Exclusion Criteria:

* Diagnosed metabolic, cardiovascular, or thyroid disorders
* Cardiac arrhythmias
* Current prescription drugs with possible cardiovascular or neurocognitive effects
* Smoking
* Known or suspected sensitivity to Rhodiola rosea
* Regular alcohol intake >12 drinks/week
* Recent musculoskeletal injury that could limit resistance-exercise testing

Ages: 18 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Load volume (kg) during 3rd set to failure at 60% 1RM | Day 7 of each 7-day period
  Participants performed bench presses and leg presses at 60% of their familiarization 1RM. On the 3rd set, they lifted to volitional failure; load volume was calculated as load (kg) × repetitions. Values after administration of low- and high-dose Rhodiola rosea were compared with those of the placebo and control groups.
Wingate anaerobic test peak power | Day 7 of each 7-day period
  Participants completed a 30-s Wingate test on a cycle ergometer; peak power (W) was recorded. Values after low- and high-dose Rhodiola rosea were compared with those of the placebo and control to assess the effects on anaerobic performance.
Executive function (Stroop Color-Word Test) | Day 7 of each 7-day period
  The paper-and-pencil Stroop Color-Word Test is administered (Word, Color, and Color-Word, 45 s each). The total number of correct responses across the three sections is recorded. Higher scores indicate better executive control.

SECONDARY OUTCOMES:
Readiness to Perform (Visual Analog Scale, 0-100 mm) | Day 7 of each 7-day period
  Participants rated six items before testing on a 0-100 mm line anchored 0 = strongly disagree (worse) and 100 = strongly agree (better): (1) I slept well last night; (2) I am looking forward to today's workout; (3) I am optimistic about my future performance; (4) I feel vigorous and energetic; (5) My appetite is great; (6) I have little muscle soreness. Scores were recorded in millimeters; higher values indicate better readiness (greater agreement).
Rating of Perceived Exertion (RPE) after resistance exercise | Day 7 of each 7-day period
  RPE is recorded 1 minute after the 3rd set of bench press and leg press using the Borg 6-20 scale. Higher values indicate greater perceived exertion.
Resting Heart Rate | Day 7 of each 7-day period
  Seated/resting heart rate measured before testing. Unit: beats per minute (bpm). Higher values indicate higher HR.
1-Minute Post-Exercise Heart Rate | Day 7 of each 7 days (1-min post-bench press; 1-min post-leg press; 1-min post-Wingate).
  Heart rate was measured 60 s after completion of each exercise bout (bench press, leg press, Wingate). Unit: beats per minute (bpm). Higher values indicate higher HR.
Resting Systolic Blood Pressure | Day 7 of each 7 days (pre-test).
  Seated/resting SBP measured before testing using an automated oscillometric device per manufacturer guidelines. Unit: mmHg. Higher values indicate higher SBP.
Resting Diastolic Blood Pressure | Day 7 of each 7 days (pre-test).
  Seated/resting DBP measured before testing using an automated oscillometric device per manufacturer guidelines. Unit: mmHg. Higher values indicate higher DBP.
1-Minute Post-Exercise Systolic Blood Pressure | Day 7 of each 7 days (1-min post-bench press; 1-min post-leg press; 1-min post-Wingate).
  SBP was measured 60 s after completion of each exercise bout (bench press, leg press, Wingate). Unit: mmHg. Higher values indicate higher SBP.
1-Minute Post-Exercise Diastolic Blood Pressure | Day 7 of each 7 days (1-min post-bench press; 1-min post-leg press; 1-min post-Wingate).
  DBP was measured 60 s after completion of each exercise bout (bench press, leg press, Wingate). Unit: mmHg. Higher values indicate higher DBP.
Adverse Events / Side-Effects-Frequency (0-5 Likert) | Day 7 of each 7 days (post-condition).
  Participants completed a side-effects questionnaire rating how often each symptom occurred using a 6-point scale (0 = none; 1 = minimal [1-2/week]; 2 = slight [3-4/week]; 3 = occasional [5-6/week]; 4 = frequent [7-8/week]; 5 = severe [≥9/week]). Symptoms queried: dizziness, headache, fast/racing heart rate, heart skipping/palpitations, shortness of breath, nervousness, blurred vision, and "any other unusual/adverse effects." Scores range 0-5 per item; higher = worse (more frequent). Each item was analyzed separately; an optional composite frequency score (item mean) was also recorded.
Adverse Events / Side-Effects-Severity (0-5 Likert) | Day 7 of each 7 days (post-condition).
  Description: Using the same questionnaire, participants rated how severe each symptom was on a 6-point scale (0 = none; 1 = minimal; 2 = slight; 3 = moderate; 4 = severe; 5 = very severe). Symptoms queried: dizziness, headache, fast/racing heart rate, heart skipping/palpitations, shortness of breath, nervousness, blurred vision, and "any other unusual/adverse effects." Scores range 0-5 per item; higher = worse (more severe). Each item was analyzed separately; an optional composite severity score (item mean) was also recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology and Nutrition Laboratory (EPNL) at Jacksonville State University, Jacksonville, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset is small, includes performance and health-related variables that may permit re-identification of participants from a single institution, and consent did not explicitly cover public data sharing.